CLINICAL TRIAL: NCT03340701
Title: Pharmacokinetics of Vaginal Progesterone in Pregnancy
Brief Title: Pharmacokinetics of Progesterone in Pregnancy
Acronym: PK-PiP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17D.559
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Progesterone
Keywords: progesterone; pharmacology; pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic study to assess plasma concentration time profile of vaginal progesterone in pregnant women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vaginal Progesterone (Other): micronized progesterone vaginal suppository 200mg
  Interventions: Drug: vaginal progesterone suppository

INTERVENTIONS:
Drug: vaginal progesterone suppository — 200mg vaginal suppository micronized progesterone

SUMMARY:
Pharmacokinetic analysis of 200mg vaginal progesterone suppository in women with singleton pregnancies between 18 0/7- 23 6/7 weeks' gestation

DETAILED DESCRIPTION:
Prospective study of 6 women with singleton pregnancies 18 0/7- 23 6/7 weeks' gestation with no prior preterm birth or short cervix who are administered a single dose of 200mg vaginal progesterone suppository. Serum progesterone levels will be drawn serially from pre-dose to 24 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old pregnant with singleton gestation 16 0/7 - 23 6/7 weeks
* pre-pregnancy BMI 20-40
* no history of prior preterm birth

Exclusion Criteria:

* history of an adverse reaction to progesterone
* contraindication to progesterone treatment including prior or active thrombus, active hepatic disease, known adverse reaction to progesterone
* medical comorbidity requiring medication including: hypertension, diabetes, substance abuse/methadone maintenance therapy, asthma, thyroid disease
* major fetal anomaly diagnosed on ultrasound or known chromosomal disorder
* multifetal gestation
* vaginal bleeding, preterm labor, premature rupture of membranes, or clinical chorioamnionitis, at the time of enrollment or on Day 1 of study
* any progesterone use of any form previously during the pregnancy
* active vaginitis
* Illicit substance use in pregnancy including cocaine, opiates, marijuana
* abnormal pap smear/+HPV on most recent pap smear
* known or suspected malignancy of the breast or genital organs
* cervical length ≤25mm

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only women, study in pregnancy
Enrollment: 6 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic model | 24 hours
  Plasma concentration time profile of vaginal progesterone in pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: Rupsa C Boelig, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Boelig RC, Zuppa AF, Kraft WK, Caritis S. Pharmacokinetics of vaginal progesterone in pregnancy. Am J Obstet Gynecol. 2019 Sep;221(3):263.e1-263.e7. doi: 10.1016/j.ajog.2019.06.019. Epub 2019 Jun 15. PMID 31211965